CLINICAL TRIAL: NCT05068414
Title: Evaluation De L'incidence Des Évènements Hémorragiques Et Ischémiques En Post-angioplastie Chez Des Patients Coronariens Anticoagulés Dans Le Cadre D'une Fibrillation Auriculaire
Brief Title: Assessment of the Incidence of Hemorrhagic and Ischemic Events in Post-angioplasty in Anticoagulated Coronary Patients with Atrial Fibrillation
Acronym: FACOREV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2020/AJ-01
Record Dates: First submitted 2021-09-27; First posted 2021-10-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation; Acute Coronary Syndrome; Thrombosis; Hemorrhage
Keywords: dual anti-platelet therapy; angioplasty
MeSH Terms: conditions — Atrial Fibrillation; Acute Coronary Syndrome; Thrombosis; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with atrial fibrillation
  Interventions: Diagnostic Test: Blood panel

INTERVENTIONS:
Diagnostic Test: Blood panel — * Thrombin generation test
  * Residual plasma concentration of dabigatran, rivaroxaban and/or apixaban (direct oral anticoagulants)
  * International Normalized Ratio (if anti-vitamin K therapy is prescribed)
  * Platelet aggregation test

SUMMARY:
Atrial fibrillation (AF) is a supraventricular arrhythmia characterized by uncoordinated and fast atrial activity, and coronary artery disease (chronic and acute coronary syndrome) is characterized by a generally atheromatous narrowing of the coronary arteries. Angioplasty is necessary to restore arterial circulation in coronary artery disease. A dual anti-aggregating therapy is then initiated in these patients in parallel with treatment of AF with anticoagulation. This triple therapy exposes the patient to an increased risk of hemorrhage. The combination of oral anticoagulation with antiplatelet inhibitor in long-term anticoagulated patients requiring stent placement has been studied in several recent trials (e.g. WOEST, PIONEER AF PCI, REDUAL PCI and AUGUSTUS). The results of these studies have formed the basis of the European recommendations of 2017 and 2020, whereby the therapeutic strategy depends on the risk of hemorrhage or ischemia. However, the hemorrhagic risk assessment factors included in the scores overlap with those for ischemic risk. It is therefore difficult to determine the predominant risk for each patient. Thus, uncertainties persist as to the optimal duration of a triple therapy and the optimal recommended dose.

In this study, the investigators aim to establish an inventory of the current practices by evaluating the incidence of hemorrhagic and ischemic events in post-angioplasty in anticoagulated coronary patients in the context of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patient on anti-coagulating therapy before or during hospitalization for atrial fibrillation
* Patient hospitalized in the cardiology ward admitted for acute or chronic coronary syndrome requiring coronary angioplasty
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is in a period of exclusion determined by a previous study
* The patient has already been included into this study
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient pregnant, parturient or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at least 18 years of age admitted for hospitalization in the cardiology department of the Nîmes Hospital for angioplasty as part of an acute or chronic coronary syndrome and being anticoagulated before or during their hospitalization for a paroxysmal, persistent or permanent atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
Incidence of at least one event from the composite clinical benefit endpoints: death, non-fatal myocardial infarction, ischemic stroke, or major bleeding defined by a Bleeding Academic Research Consortium (BARC) score ≥2 | Month 12
  Number of patients

SECONDARY OUTCOMES:
Incidence of at least one event from the composite clinical benefit endpoints: death, non-fatal myocardial infarction, ischemic stroke, or major bleeding defined by a Bleeding Academic Research Consortium (BARC) score ≥2 | Month 1
  Number of patients
Incidence of at least one event from the composite clinical benefit endpoints: death, non-fatal myocardial infarction, ischemic stroke, or major bleeding defined by a Bleeding Academic Research Consortium (BARC) score ≥2 | Month 6
  Number of patients
Occurrence of stent thrombosis | Month 1
  Number of patients
Occurrence of stent thrombosis | Month 6
  Number of patients
Occurrence of stent thrombosis | Month 12
  Number of patients
Occurrence of stroke | Month 1
  Number of patients
Occurrence of stroke | Month 6
  Number of patients
Occurrence of stroke | Month 12
  Number of patients
Occurrence of myocardial infarction | Month 1
  Number of patients
Occurrence of myocardial infarction | Month 6
  Number of patients
Occurrence of myocardial infarction | Month 12
  Number of patients
Occurrence of death from any cause | Month 1
  Number of patients
Occurrence of death from any cause | Month 6
  Number of patients
Occurrence of death from any cause | Month 12
  Number of patients
Occurrence of revascularization of the target lesion without death | Month 1
  Number of patients
Occurrence of revascularization of the target lesion without death | Month 6
  Number of patients
Occurrence of revascularization of the target lesion without death | Month 12
  Number of patients
Occurrence of peripheral embolism | Month 1
  Number of patients
Occurrence of peripheral embolism | Month 6
  Number of patients
Occurrence of peripheral embolism | Month 12
  Number of patients
Stroke risk | Month 1
  ABCD2 score
Stroke risk | Month 6
  ABCD2 score
Stroke risk | Month 12
  ABCD2 score
Intrinsic imputability of transient ischemic attack | Month 12
  According to French pharmacovigilance scale from I0 (incompatible) to I4 (very likely)
Extrinsic imputability of transient ischemic attack | Month 12
  According to French pharmacovigilance scale from B0 (Effect appearing quite new after exhaustive research) to B3 (notable effect)
Intrinsic imputability of hemorrhagic eccent | Month 12
  According to French pharmacovigilance scale from I0 (incompatible) to I4 (very likely)
Extrinsic imputability of hemorrhagic eccent | Month 12
  According to French pharmacovigilance scale from B0 (Effect appearing quite new after exhaustive research) to B3 (notable effect)
Bleeding Academic Research Consortium Score | Month 1
  Classified according to subcategories; 1-5; 2-5; or 3-5
Bleeding Academic Research Consortium Score | Month 6
  Classified according to subcategories; 1-5; 2-5; or 3-5
Bleeding Academic Research Consortium Score | Month 12
  Classified according to subcategories; 1-5; 2-5; or 3-5
Number of anti-platelet aggregations taken | Month 1
  Number
Number of anti-platelet aggregations taken | Month 6
  Number
Number of anti-platelet aggregations taken | Month 12
  Number
Anatomical Therapeutic Chemical class of anti-platelet aggregation and the anticoagulants | Month 1
Anatomical Therapeutic Chemical class of anti-platelet aggregation and the anticoagulants | Month 6
Anatomical Therapeutic Chemical class of anti-platelet aggregation and the anticoagulants | Month 12
Duration of triple therapy | Month 1
Duration of triple therapy | Month 6
Duration of triple therapy | Month 12
Dose of anti-platelet aggregation and the anticoagulants | Month 1
Dose of anti-platelet aggregation and the anticoagulants | Month 6
Dose of anti-platelet aggregation and the anticoagulants | Month 12
Global drug compliance | Month 1
  Girerd score where 0 = good observance, 1/2 = slight observance problems, 3+ = poor observance
Global drug compliance | Month 6
  Girerd score where 0 = good observance, 1/2 = slight observance problems, 3+ = poor observance
Global drug compliance | Month 12
  Girerd score where 0 = good observance, 1/2 = slight observance problems, 3+ = poor observance
Compliance with antiplatelet and anticoagulant therapy | Month 1
  Girerd score specific to anticoagulation/antiplatelet: where 0 = good observance, 1/2 = slight observance problems, 2.5+ = poor observance
Compliance with antiplatelet and anticoagulant therapy | Month 6
  Girerd score specific to anticoagulation/antiplatelet: where 0 = good observance, 1/2 = slight observance problems, 2.5+ = poor observance
Compliance with antiplatelet and anticoagulant therapy | Month 12
  Girerd score specific to anticoagulation/antiplatelet: where 0 = good observance, 1/2 = slight observance problems, 2.5+ = poor observance
Thrombin generation test | Inclusion
  Kinetic fluorimetry curve, (ST Genesia® analyzer)
Thrombin generation test | Month 6
  Kinetic fluorimetry curve, (ST Genesia® analyzer)
Thrombin generation test | Month 12
  Kinetic fluorimetry curve, (ST Genesia® analyzer)
Residual plasma concentration of direct oral anticoagulants (dabigatran, rivaroxaban and apixaban) | Inclusion
  Measured with STA-R® Plus
Residual plasma concentration of direct oral anticoagulants (dabigatran, rivaroxaban and apixaban) | Month 6
  Measured with STA-R® Plus
Residual plasma concentration of direct oral anticoagulants (dabigatran, rivaroxaban and apixaban) | Month 12
  Measured with STA-R® Plus
International Normalized Ratio (INR) for patients under if anti-vitamin K therapy | Inclusion
  Measured with STA-R® Plus
International Normalized Ratio (INR) for patients under if anti-vitamin K therapy | Month 6
  Measured with STA-R® Plus
International Normalized Ratio (INR) for patients under if anti-vitamin K therapy | Month 12
  Measured with STA-R® Plus
D-dimers level | Month 1
  D-Dimer Exclusion assay
D-dimers level | Month 6
  D-Dimer Exclusion assay
D-dimers level | Month 12
  D-Dimer Exclusion assay
Fibrin monomers level | Month 1
  STA-Liatest FM
Fibrin monomers level | Month 6
  STA-Liatest FM
Fibrin monomers level | Month 12
  STA-Liatest FM
Platelet aggregation test | Inclusion
  Platelet inhibition under aspirin and/or P2Y12 inhibitor
Platelet aggregation test | Month 6
  Platelet inhibition under aspirin and/or P2Y12 inhibitor
Platelet aggregation test | Month 12
  Platelet inhibition under aspirin and/or P2Y12 inhibitor
Association between ischemic an/ord hemorrhagic events and adherence to antiplatelet therapy and anticoagulant medication initiated after stent placement | Month 12
  Rate
Concordance rate between the drug compliance score and the biological assessment | Inclusion
Concordance rate between the drug compliance score and the biological assessment | Month 6
Concordance rate between the drug compliance score and the biological assessment | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Alexia Janes, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No